CLINICAL TRIAL: NCT00278863
Title: Randomized Multicenter Phase II Trial of Capecitabine Versus S-1 as First-line Treatment in Elderly Patients With Advanced or Recurrent Unresectable Gastric Cancer
Brief Title: Capecitabine Versus S-1 in Elderly Advanced Gastric Cancer (AGC): Randomized Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC-ONCGI-0415
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-01

CONDITIONS: Gastric Cancer
Keywords: Stomach cancer; Palliative chemotherapy; Capecitabine; S-1
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-1 (Active Comparator)
  Interventions: Drug: S-1
- Capecitabine (Active Comparator)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: S-1
  Arms: S-1
Drug: Capecitabine
  Arms: Capecitabine

SUMMARY:
A significant proportion of advanced gastric cancer (AGC) occurs in individuals 65 years of age and older. In addition, patient delay in seeking care for symptoms results in diagnosis at a more advanced stage than that seen in younger individuals. However, clinical trials on gastric cancer rarely have been available to the elderly. Recently oral 5-FU pro-drugs, which have been reported to have clinically significant response rates and survival with mild or negligible toxicities, have been widely used for the patients with AGC. However, few studies have been conducted in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven gastric or gastroesophageal junction adenocarcinoma
* Metastatic or recurrent unresectable disease
* Measurable lesions (according to Response Evaluation Criteria in Solid Tumors [RECIST])
* Age: 65-85 years old
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2
* Adequate bone marrow function: absolute neutrophile counts(ANC) ≥ 1,500/ul, platelet count ≥ 100,000/ul, hemoglobin ≥ 9 g/dl)
* Adequate renal function (serum creatinine≤ 1.5)
* Adequate liver function (serum bilirubin ≤ 2 x upper limits of normal [UNL], aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x UNL)
* No prior chemotherapy (but adjuvant chemotherapy completed at least 1 year prior to study treatment is allowed with the exception of capecitabine or S-1) Written informed consent was signed by the patient

Exclusion Criteria:

* Previous palliative chemotherapy
* Known allergy to study drugs
* CNS metastasis
* Significant medical comorbidities
* Active ongoing infection which antibiotic treatment is needed.
* Previous ( within 5 years) history of other malignancy except cured non-malignant skin cancer and uterine cervical cancer in situ.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Actual)
Dates: Start 2004-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (9):
- South Korea (9):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Pyeongchon, Gyeonggido
  - Kyung Pook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Gacheon Medical School Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Seoul Samsung Medical Center, Seoul
  - Ulsan University Hospital, Ulsan

RESULTS

PARTICIPANT FLOW:
Groups:
- S-1 for 2 Week on/1 Week Off: S-1 was given orally two times daily for 28 days, followed by 14 days' rest. Three dosage levels of S-1 were defined according to body surface area (BSA) as follows: BSA less than 1.25 m2, 40mg two times daily; BSA, 1.25 to 1.5 m2, 50 mg, two times daily; and BSA more than 1.5 m2, 60 mg two times daily.
- Capecitabine 2 Weeks on/1 Week Off: Capecitabine 2500 mg square meter was administered orally in two divided doses daily on days 1-14 of a 21-day cycle.
Period: Overall Study
Arm/Group | S-1 for 2 Week on/1 Week Off | Capecitabine 2 Weeks on/1 Week Off
Started | 49 | 47
Completed | 44 | 45
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- S-1 for 2 Weeks on/1 Week Off: S-1 was given orally two times daily for 28 days, followed by 14 days' rest. Three dosage levels of S-1 were defined according to body surface area (BSA) as follows: BSA less than 1.25 m2, 40mg two times daily; BSA, 1.25 to 1.5 m2, 50 mg, two times daily; and BSA more than 1.5 m2, 60 mg two times daily.
- Total: Total of all reporting groups
Arm/Group | S-1 for 2 Weeks on/1 Week Off | Capecitabine 2 Weeks on/1 Week Off | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Customized [Median (Full Range); unit: years]
  Age_median | 71 [65 to 82] | 71 [66 to 88] | 71 [65 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 24
  Male | 37 | 30 | 67
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 45 | 46 | 91

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Progressive disease (PD), >20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD), Insufficient change to qualify for PR or PD
  Response rate is defined as the proportion of patients who showed OR.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | S-1 for 2 Week on/1 Week Off | Capecitabine 2 Weeks on/1 Week Off
Number analyzed (Participants) | 45 | 44
percentage of participants | 28.9 [15.6 to 42.1] | 26.1 [13.4 to 38.8]

2. Secondary Outcome: Number of Patients With Adverse Events
Description: Per National Cancer Institute Common Toxicity Criteria Version 2.0, up to 2 years
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | S-1 for 2 Week on/1 Week Off | Capecitabine 2 Weeks on/1 Week Off
Number analyzed (Participants) | 42 | 44
participants | 42 | 44

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | S-1 for 2 Week on/1 Week Off | Capecitabine 2 Weeks on/1 Week Off
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/44
Other Adverse Events (participants affected / at risk) | 42/42 | 44/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S-1 for 2 Week on/1 Week Off (N=42) | Capecitabine 2 Weeks on/1 Week Off (N=44)
Anemia (Blood and lymphatic system disorders) | 37 | 39
Leukopenia (Blood and lymphatic system disorders) | 14 | 10
Neutropenia (Blood and lymphatic system disorders) | 10 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 12
Asthenia (General disorders) | 34 | 34
Anorexia (Gastrointestinal disorders) | 31 | 38
Nausea (Gastrointestinal disorders) | 23 | 22
Vomiting (Gastrointestinal disorders) | 10 | 10
Abdominal pain (Gastrointestinal disorders) | 20 | 19
Stomatitis (Gastrointestinal disorders) | 9 | 24
Diarrhea (Gastrointestinal disorders) | 13 | 16
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 7 | 26
Hyperbilirubinemia (Hepatobiliary disorders) | 13 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No